CLINICAL TRIAL: NCT05995626
Title: Hyaluronidase Via Laser-Assisted Drug Delivery for the Treatment of Scleroderma-induced Microstomia
Brief Title: Hyaluronidase Via LADD Scleroderma-induced Microstomia
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0210-23-FB
Record Dates: First submitted 2023-08-08; First posted 2023-08-16 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Microstomia; Scleroderma
MeSH Terms: conditions — Microstomia; Scleroderma, Diffuse | interventions — Hyaluronoglucosaminidase; Chondroitinases and Chondroitin Lyases; Lasers, Gas

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Ablative CO2 laser, and intradermal hyaluronidase, via laser-assisted drug delivery (Experimental): Uncover a safe, efficacious, and tolerable alternate treatment modality for scleroderma-induced microstomia. Evaluate disease severity and participant quality of life before and after alternative treatment.
  Interventions: Drug: Hyaluronidase; Device: CO2 laser

INTERVENTIONS:
Drug: Hyaluronidase — Hyaluronidase injection is used during fluid administration under the skin to help achieve hydration, to increase the dispersion and absorption of other injected drugs, or during some types of urography (imaging of the urinary tract) to help improve resorption of drugs used during the procedure.
  Other Names: Vitrase
Device: CO2 laser — CO2 lasers use an aiming beam to see where the treatment beam will impact the focus tissue, which will then be cleanly incised. The CO2 lasers have greater precision for laser surgery and have more flexibility in tip sizes and protocols.

SUMMARY:
Two treatment methods, ablative carbon dioxide (CO2) laser and intradermal hyaluronidase, will be combined to maximize the beneficial potential of each. Laser-assisted drug delivery (LADD) has been shown to be effective for the administration of medications in diverse skin diseases but not previously reported for the treatment of scleroderma-induced microstomia. By using this laser technique, the investigator can reduce the pain of typical hyaluronidase injections and reap the therapeutic benefit of the laser treatment itself. The investigator's goal is to create greater mouth mobility for chewing and speaking as well as improved oral hygiene, self-esteem, and overall quality of life. Each participant will undergo three separate laser sessions at 4 to 8-week intervals. Participants will also complete a follow-up visit three months after the last laser session to evaluate the response.

DETAILED DESCRIPTION:
In this study, the investigator will combine two treatment modalities, ablative carbon dioxide (CO2) laser, and intradermal hyaluronidase, via laser-assisted drug delivery. The goal is to maximize the therapeutic potential of each of these interventions by combining them. Laser-assisted drug delivery (LADD) has been shown to be an effective modality for the administration of medications in diverse cutaneous diseases but has not been previously reported for the treatment of scleroderma-induced microstomia. By using an ablative fractional CO2 laser, the investigator can facilitate both the intradermal administration of hyaluronidase and the therapeutic benefit of the laser treatment itself. LADD of hyaluronidase has the additional advantage of being less painful and likely better tolerated than intradermal hyaluronidase injections, which typically require painful infraorbital and mental nerve blocks. The goal is to provide participants with a novel, effective, and less painful option for the treatment of scleroderma-induced microstomia, leading to greater mouth mobility for mastication and phonation as well as improved oral hygiene, self-esteem, and overall quality of life.

Ten participants with scleroderma-induced microstomia will be selected primarily from the scleroderma patient population at University of Nebraska Medical Center (UNMC) Dermatology as well as from a local non-profit scleroderma support group. Each participant will undergo three separate laser sessions. On each occasion, investigators will treat the perioral area with 200 units of hyaluronidase, administered via LADD using an ablative fractional CO2 laser. These appointments will be scheduled at 4 to 8-week intervals, depending on the participant's tolerance to laser therapy and availability. Participants will also complete a non-procedural follow-up visit three months after the last laser session to evaluate for a sustained response.

ELIGIBILITY:
Inclusion Criteria:

* Patient at the Lauritzen Outpatient Clinic or Westroads Clinic, Dept Dermatology
* Diagnosed with scleroderma-induced microstomia
* Capable and willing to participate
* Free of medical conditions that will interfere with successful completion of the study, such as severe dementia or seizure disorder
* Aged 19 or older

Exclusion Criteria:

* Pregnant and breastfeeding women
* 18 years old or younger
* Infections or inflammation in or near the area of treatment
* Prior treatment with hyaluronidase, LADD or ablative CO2 laser treatment, or a history of adverse reactions to the treatments

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-09-24 (Actual); Study Completion 2024-09-24 (Actual)

PRIMARY OUTCOMES:
Difference in Interincisal Distance | 6 months
  The aim is to increase interincisal distance. Measurements will be collected before and after every treatment and on follow-up visit.

SECONDARY OUTCOMES:
Difference in Mouth Handicap In Systemic Sclerosis Score | Baseline and 6 months
  Mouth handicap in systemic sclerosis score is a subjective measurement of the impact of microstomia in scleroderma patients. It is answered according to the five-point Likert system: 0: Never, 1: Rarely, 2: Sometimes, 3: Frequently, 4: Always. The higher the total score, the higher the severity of the problem. The aim is to evaluate the score difference before and after the completion of treatment.
Differences in Inter-labial and Inter-commissural Distance | Baseline and 6 months
  The aim is to increase both distances. These measurements will be collected before and after every treatment and on follow-up visit.
Quality of life RAND 36-item Health Survey 1.0 | Baseline and 6 months
  The aim is to assess the impact of our treatment modality on quality of life. Participants will fill out a questionnaire before the start and after the completion of treatment.
Treatment Satisfaction | 6 months
  Participant's satisfaction with treatment will be measured with a Likert Scale, 1 = very dissatisfied and 5 = very satisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah L Lonowski, MD, Principal Investigator — University of Nebraska
Locations (2):
- United States (2):
  - University of Nebraska Medical Center, Lauritzen Outpatient Center, Omaha, Nebraska
  - Nebraska Medicine, Dermatology Westroads, Omaha, Nebraska

IPD SHARING:
Plan to Share IPD: No